CLINICAL TRIAL: NCT07258940
Title: A 1-year Prospective Multicenter Clinical Investigation to Assess Safety, Performance and Clinical Benefits of the NobelZygoma TiUltra Implant System in the Rehabilitation of Severely Atrophic Maxillae
Brief Title: NobelZygoma TiUltra Implant System Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-197
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Edentulous Maxilla; Maxillary Bone Loss; Atrophic Maxilla
Keywords: "zygomatic implants"; "zygoma implants"
MeSH Terms: conditions — Atrophic Maxilla

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, multicenter, single cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NobelZygoma TiUltra implant system in the rehabilitation of severely atrophic maxillae (Other): Participant will receive zygomatic implant treatment for the rehabilitation of severely atrophic maxilla. The treatment will be performed as per standard-of-care and participant's anatomic conditions. The NobelZygoma TiUltra implant and Multi-unit Abutment Xeal Zygoma will be used in all study participants.
  Interventions: Device: NobelZygoma™ 0° CC TiUltra™implant ; NobelZygoma™ 45° Ext Hex TiUltra™ implant; Device: Multi-Unit Abutment Xeal Zygoma Ext Hex RP; 17° Multi-Unit Abutment Xeal Zygoma Ext Hex RP; 45° Multi.Unit Abutment Xeal Zygoma CC RP; 60° Multi-Unit Abutment Xeal Zygoma CC RP

INTERVENTIONS:
Device: NobelZygoma™ 0° CC TiUltra™implant ; NobelZygoma™ 45° Ext Hex TiUltra™ implant — All participants will receive NobelZygoma TiUltra implant and Multi-unit Abutment Xeal as part of the implant/prosthetic zygomatic rehabilitation procedure. Implants and abutments will be selected as per surgeon preference and participant's need. Radiological exam will be performed at pre-treatment and 12-months follow-up. Patients will be followed-up after placement of implant at 10-days, 6-months and 12-months follow-up. At 12-months a standardized clinical and radiological criteria (using the SNOT-22 and Lund-Mackay respectively) will be used to describe and quantify the occurrence of maxillary sinusitis across all study centers for the sinusitis diagnose.
Device: Multi-Unit Abutment Xeal Zygoma Ext Hex RP; 17° Multi-Unit Abutment Xeal Zygoma Ext Hex RP; 45° Multi.Unit Abutment Xeal Zygoma CC RP; 60° Multi-Unit Abutment Xeal Zygoma CC RP — All participants will receive NobelZygoma TiUltra implant and Multi-unit Abutment Xeal as part of the implant/prosthetic zygomatic rehabilitation procedure. Implants and abutments will be selected as per surgeon preference and participant's need. Radiological exam will be performed at pre-treatment and 12-months follow-up. Patients will be followed-up after placement of implant at 10-days, 6-months and 12-months follow-up. At 12-months a standardized clinical and radiological criteria (using the SNOT-22 and Lund-Mackay respectively) will be used to describe and quantify the occurrence of maxillary sinusitis across all study centers for the sinusitis diagnose

SUMMARY:
The goal of this prospective study is to assess short term (12-months) clinical outcomes of NobelZygoma TiUltra implants and Multi-unit Abutment Xeal in the rehabilitation of participants with severely atrophic maxilla treated with zygomatic dental implant procedure. The main goal is to assess the sinusitis occurrence at 12-months after implant insertion. Other objectives are to assess: soft tissue health; biological and technical complication; patient's experience, outcomes (sinonasal symptoms and oral health-related quality of life) and satisfaction; clinician's experience with handling of device and satisfaction; implant, abutment and prosthetic survival and adverse events.

Participants will be asked to complete questionnaires at pretreatment visit, postoperative visit, and after 6-months and 12-months of implant insertion. At 12-months a radiological exam (CBCT) will be asked for the participant for the evaluation of the radiological condition of the maxillary sinus.

DETAILED DESCRIPTION:
This is a prospective, interventional, multicenter study that is planned to include 9 sites and 85 participants with severely atrophic maxilla (characterized by class V-VI according to the Cawood and Howell's classification). Participants will be consecutively enrolled upon providing informed consent and meeting all of the inclusion and none of the exclusion criteria (details in eligibility section). Zygomatic implant procedure will be performed as per clinician standard of care and participant's anatomy. Both hybrid and quad zygoma techniques, as well as any implant trajectory can be used in the study (e.g. intra-sinus; extra-sinus; sinus slot). Enrolled participants will be treated with NobelZygoma TiUltra implants and respective abutments in accordance with the IFU. All zygomatic implants will be immediately loaded.

The study is designed to describe and quantify the occurrence of maxillary sinusitis in participants treated with NobelZygoma TiUltra implants and Multi-unit Abutments Xeal Zygoma.

The working assumption is that the incidence of sinusitis can be reliably measured at 12 months using standardized clinical (SNOT-22) and radiological (Lund-Mackay) criteria in participants rehabilitated with this treatment approach The primary endpoint of this clinical investigation is the specificity of diagnosis of maxillary sinusitis at 12-months post-implant placement using a combination of clinical and radiological evaluation, using SNOT-22 questionnaire and LM (Lund-Mackay) scoring system for the clinical and CBCT analysis respectively. Other endpoint and parameters will be described in Outcome measures section.

All included participants will be followed for 12-months post-implant placement to assess the safety, performance, and clinical benefits of TiUltra-surfaced zygomatic implants and Mulit-unit Abutment Xeal Zygoma. Possible dropouts and withdrawals, as well as possible adverse events, will be monitored during the entire investigation period.

Each participant will be assigned a participant ID to maintain the confidentiality of the collected data, which will be recorded in the dedicated eCRF. The eCRF system meets EU GDPR requirements for safe data handling. The data will be processed by the eCRF provider for storage purposes and further processed and analyzed by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Participant has signed the informed consent form (ICF).
* Participant aged ≥ 18 years at the time of treatment.
* Medical and anatomical conditions are in accordance with the applicable IFU.
* Participant with a severely atrophic maxilla classified as Cawood and Howell class V or VI
* Suitable for immediate loading.

Exclusion Criteria:

* Presence of acute or chronic maxillary sinusitis.
* Zygomatic bone pathologies including tumors, infections, or congenital abnormalities
* History of recurrent sinusitis (≥ 4 occurrences/year)
* Pre-operative LM score of ≥ 1
* Uncontrolled systemic disorders including poorly controlled hypertension, uncontrolled diabetes, cardiovascular disease.
* Active malignancy or currently undergoing oncological treatment.
* History of severe maxillary jaw injury or maxillofacial trauma.
* Moderate and heavy smokers (defined as > 5 cigarettes a day).
* Severe bruxism or dysfunctional tendencies
* Previous oro-maxillofacial radiotherapy.
* Use of bisphosphonates.
* Pregnant or lactating women
* Implant loaded > 1 week of zygomatic implant placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Maxillary sinusitis at 12-months post-implant placement | At 12-months follow-up of zygomatic implant insertion
  The diagnosis of maxillary sinusitis is based on the following criteria:
  A positive clinical diagnosis is made when all of the following criteria from SNOT-22 are met simultaneously:
  1. The participant reports at least two clinical symptoms, one of which must be either: nasal blockage/obstruction/congestion, or nasal discharge (anterior or posterior nasal drip). Additional symptoms may include: facial pain or pressure, reduction or loss of smell.
  2. There is a clinically significant worsening in symptoms, demonstrated by a ≥12-point increase in the total SNOT-22 score from baseline (pre-treatment).
  3. If the participant exhibits partial symptoms or if the diagnosis remains uncertain, the Principal Investigator (PI) will refer the participant to an ENT specialist for further evaluation.

SECONDARY OUTCOMES:
PREMs | At pre-treatment; and after 10 days, 6- and 12-months of zygomatic implant placement
  Evaluate patient reported experience measures (PREMs) from pre-treatment to 12-month follow-up using Likert scale
Pain assessment | 10 days after zygomatic implant placement
  Assess patient reported pain at postoperative visit using VAS scale (from 0 (no pain) to 100 (worst pain possible)
Patient satisfaction | 10 days, 6-months and 12-months after zygomatic implant placement
  Assess patient satisfaction with function and esthetics using VAS scale (from 0 - not satisfied to 100 fully satisfied
OHIP-21 | At pre-treatment and after 10 days, 6-months and 12-months of zygomatic implant placement
  Evaluate oral health-related quality of life using OHIP-21 questionnaire from pre-treatment to 12-month follow-up.
Keratinized mucosa status | At 6-months and 12-months follow-up of zygomatic implant placement
  Keratinized mucosa status will be evaluated per zygomatic implant, without the prosthesis in place, and using the following score:
  0 =No keratinized mucosa around the implant
  1. =Mucosa surrounding the implant is partially keratinized
  2. = The entire mucosa surrounding the implant is keratinized
Modified Bleeding Index (mBI) | At 6- and 12-months follow-up of zygomatic implant placement
  The mBI will be evaluated at zygomatic implant level, without the prosthesis in place, using the following score system:
  0=No bleeding when a periodontal probe is passed along the gingival margin adjacent to the implant
  1. Isolated bleeding spots visible.
  2. Blood forms a confluent red line on the margin.
  3. Heavy or profuse bleeding.
Biological | From implant placement until12-months after implant placement
  Biological complications will be recorded
Adverse Events | From implant placement until 12-months after implant placement
  All adverse events (AEs), serious adverse events (SAEs), adverse device effects (ADEs), serious adverse device effects (SADEs), device deficiencies (DDs), and unanticipated serious adverse device effects (USADEs) will be recorded from implant placement to the 12-month follow-up.
Implant survival rate | From time of placement to 12-months follow-up
  Evaluate implant survival rate from time of placement to 12-months follow-up
Abutment survival rate | From implant placement to 12-months follow-up
  Evaluate abutment survival rate from implant placement to 12-months follow-up
Clinician satisfaction - handling of device | After 10-days of zygomatic implant placement
  To evaluate clinician's satisfaction with handling of the device using a VAS scale (from 0-not satisfied to 100-fully satisfied)
Clinician satisfaction - function and esthetic | At 6-months and 12-months follow-up of zygomatic implant placement
  To evaluate clinician's satisfaction with function and esthetics (using VAS scale 0-not satisfied and 100-fully satisfied)
Technical complications | From zygomatic implant placement until 12.months follow-up
  All technical complications will be recorded

OTHER OUTCOMES:
Prosthetic survival | From placement until 12-months follow-up
  To evaluate prosthetic survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Bednarek, Study Director — Nobel Biocare
Locations (2):
- Universitiy of Verona, Unit of Stomatology and Maxillo-Facial Surgery, Verona, Italy
- Hirslanden Medical Center, Aarau, Switzerland

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. As per data protection regulation in EU participant's identity should be kept confidential. As per informed consent and GDPR consent, participant is informed that their data will be securely stored in EDC system in EU and analyzed in Switzerland by the sponsor. As per EU and Switzerland data protection regulations, access to participant's data should only be given for the sponsor, regulatory authorities and ethic committee members. Study results will be disseminated through peer-reviewed publications and/or conference presentations. Summary results will be shared (e.g. via publication or posting results in ClinicalTrials.gov)

REFERENCES:
- [Background] Yalcin M, Can S, Akbas M, Dergin G, Garip H, Aydil BA, Varol A. Retrospective Analysis of Zygomatic Implants for Maxillary Prosthetic Rehabilitation. Int J Oral Maxillofac Implants. 2020 Jul/Aug;35(4):750-756. doi: 10.11607/jomi.8196. PMID 32724927
- [Background] Hirsch JM, Ohrnell LO, Henry PJ, Andreasson L, Branemark PI, Chiapasco M, Gynther G, Finne K, Higuchi KW, Isaksson S, Kahnberg KE, Malevez C, Neukam FW, Sevetz E, Urgell JP, Widmark G, Bolind P. A clinical evaluation of the Zygoma fixture: one year of follow-up at 16 clinics. J Oral Maxillofac Surg. 2004 Sep;62(9 Suppl 2):22-9. doi: 10.1016/j.joms.2004.06.030. PMID 15332178
- [Background] Davo R, Bankauskas S, Laurincikas R, Kocyigit ID, Mate Sanchez de Val JE. Clinical Performance of Zygomatic Implants-Retrospective Multicenter Study. J Clin Med. 2020 Feb 9;9(2):480. doi: 10.3390/jcm9020480. PMID 32050501
- [Background] Borgonovo A, Grandi T, Vassallo S, Signorini L. Extrasinus Zygomatic Implants for the Immediate Rehabilitation of the Atrophic Maxilla: 1-Year Postloading Results From a Multicenter Prospective Cohort Study. J Oral Maxillofac Surg. 2021 Feb;79(2):356-365. doi: 10.1016/j.joms.2020.10.003. Epub 2020 Oct 13. PMID 33160924
- [Background] Aparicio C, Polido WD, Chow J, Davo R, Al-Nawas B. Round and flat zygomatic implants: effectiveness after a 1-year follow-up non-interventional study. Int J Implant Dent. 2022 Apr 1;8(1):13. doi: 10.1186/s40729-022-00412-8. PMID 35359196